CLINICAL TRIAL: NCT00079898
Title: Modulatory Effect of Acupuncture on Human Brain Activity
Brief Title: Effect of Acupuncture on Human Brain Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: R21AT000978-01A1 (NIH)
Record Dates: First submitted 2004-03-18; First posted 2004-03-19 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Healthy
MeSH Terms: interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
The purpose of this study is to use brain imaging technology to examine the way acupuncture affects brain function.

DETAILED DESCRIPTION:
Acupuncture is emerging as an important procedure in complementary medicine. Its mechanism of action remains unclear, but research suggests that its effects are mediated through a widely connected network that is involved in the regulation of mood, behavior, and function of physiological systems. This study will use functional magnetic resonance imaging (fMRI) to monitor the effects of manual acupuncture on the brain function of study participants.

Participants in this study will undergo acupuncture one needle at a time. Researchers will then ask participants questions about how they feel and will compare the sensations reported by participants to their images of brain response.

ELIGIBILITY:
Inclusion Criteria:

* In good physical health

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-07; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Hui, MD, Principal Investigator — Massachusetts General Hospital

REFERENCES:
- [Background] Hui KK, Liu J, Makris N, Gollub RL, Chen AJ, Moore CI, Kennedy DN, Rosen BR, Kwong KK. Acupuncture modulates the limbic system and subcortical gray structures of the human brain: evidence from fMRI studies in normal subjects. Hum Brain Mapp. 2000;9(1):13-25. doi: 10.1002/(sici)1097-0193(2000)9:13.0.co;2-f. PMID 10643726